CLINICAL TRIAL: NCT02031237
Title: MRI Study of Changes in Blood-Brain/Tumor-Barrier Permeability in Patients With Brain Metastases During and After Radiotherapy
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2005.003; HUM00043426 (Other: University of Michigan)
Record Dates: First submitted 2013-11-13; First posted 2014-01-09 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Imaging; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Stereotactic Radiosurgery (SRS): Patients with brain metastases receiving single fraction Stereotactic Radiosurgery (SRS). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed approximately 1-2 weeks prior to SRS, and 1-2 weeks and 1 month after SRS. The MRI scan will include a routine clinical MRI series.
  Interventions: Radiation: Single Fraction Stereotactic Radiosurgery (SRS); Device: Magnetic Resonance Imaging (MRI) Assessments
- Whole Brain Radiation Therapy: Patients with brain metastases receiving fractionated (spread out over time) Whole Brain Radiation Therapy (WBRT). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed approximately 1-2 weeks prior to RT, at the end of RT and 1 month after RT. The MRI scan will include a routine clinical MRI series.
  Interventions: Radiation: Fractionated Whole Brain Radiation Therapy (WBRT); Device: Magnetic Resonance Imaging (MRI) Assessments
- Stereotactic Radiation Therapy: Patients with brain metastases receiving fractionated (spread out over time) Stereotactic Radiation Therapy (FSRT). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed approximately 1-2 weeks prior to FSRT, during the last week of RT but before the last fraction and 1 month after RT. The MRI scan will include a routine clinical MRI series.
  Interventions: Radiation: Fractionated Stereotactic Radiation Therapy (FSRT); Device: Magnetic Resonance Imaging (MRI) Assessments

INTERVENTIONS:
Radiation: Single Fraction Stereotactic Radiosurgery (SRS) — Intervention will not be assigned by the investigator. Treatment determination will be made prior to study enrollment.
  Groups: Stereotactic Radiosurgery (SRS)
Radiation: Fractionated Whole Brain Radiation Therapy (WBRT) — Intervention will not be assigned by the investigator. Treatment determination will be made prior to study enrollment.
  Groups: Whole Brain Radiation Therapy
Radiation: Fractionated Stereotactic Radiation Therapy (FSRT) — Intervention will not be assigned by the investigator. Treatment determination will be made prior to study enrollment.
  Groups: Stereotactic Radiation Therapy
Device: Magnetic Resonance Imaging (MRI) Assessments — MRI scans will include a routine clinical MRI series.

SUMMARY:
This study aims to assess changes in vascular permeability in the brain tumor, and in the surrounding brain, due to radiation therapy, using Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological confirmed malignancy and presence of intraparenchymal brain metastases
* Patients are treated by WBRT, SRS, or FSRT
* Age greater than or equal to 18 years
* A life expectancy of greater than or equal to 8 weeks
* Karnofsky performance status (an assessment of general well being and ability to do activities of daily living; scale ranges from 0 to 100 where 100 is perfect health) greater than or equal to 60
* Informed consent with signed study-specific informed consent form

Exclusion Criteria:

* Major medical or psychiatric illness, which, in the investigator's opinion, will prevent completion of the protocol
* Patients with lepto-meningeal metastases documented by Magnetic Resonance Imagine (MRI), Computed Tomography (CT), or Cerebrospinal Fluid (CSF) evaluation
* For patients that will undergo Whole Brain Radiation Therapy (WBRT), previous WBRT is not allowed. Patients who have had brain metastases managed by Stereotactic Radiosurgery (SRS), Fractionated Stereotactic Radiation Therapy (FSRT), or surgery are eligible
* For patients that will undergo Stereotactic Radiosurgery (SRS), previous Whole Brain Radiation Therapy (WBRT) within 5 months prior to study entry is not allowed. Prior Stereotactic Radiosurgery (SRS), Fractionated Stereotactic Radiation Therapy (FSRT), or surgery is allowed if current treatment will be for a lesion(s) not previously treated.
* For patients that will undergo Fractionated Stereotactic Radiation Therapy (FSRT), previous Whole Brain Radiation Therapy (WBRT) within 5 months prior to study entry is not allowed. Prior Stereotactic Radiosurgery (SRS), Fractionated Stereotactic Radiation Therapy (FSRT), or surgery is allowed if current treatment will be for a lesion(s) not previously treated.
* Patients unable to undergo or tolerate MRI scans (presence of cardiac pacemaker, implanted cardiac defibrillator, aneurysm clips, etc).
* Patients should have no contraindications to having a contrast enhanced Magnetic Resonance Imaging (MRI) scan. These contraindications will be assessed at the time of enrollment using the guidelines set up and in clinical use by the University of Michigan.
* Women who are pregnant are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain metastasis receiving radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2005-04; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Cao, Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only participants enrolled onto SRS and Whole Brain Radiation Therapy arms were evaluated for the study outcomes.
Groups:
- Stereotactic Radiosurgery (SRS): Patients with brain metastases receiving single fraction Stereotactic Radiosurgery (SRS). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed approximately 1-2 weeks prior to SRS, and 1-2 weeks and 1 month after SRS. The MRI scan will include a routine clinical MRI series.
  Single Fraction Stereotactic Radiosurgery (SRS): Intervention will not be assigned by the investigator. Treatment determination will be made prior to study enrollment.
  Magnetic Resonance Imaging (MRI) Assessments: MRI scans will include a routine clinical MRI series.
- Whole Brain Radiation Therapy: Patients with brain metastases receiving fractionated (spread out over time) Whole Brain Radiation Therapy (WBRT). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed approximately 1-2 weeks prior to RT, at the end of RT and 1 month after RT. The MRI scan will include a routine clinical MRI series.
  Fractionated Whole Brain Radiation Therapy (WBRT): Intervention will not be assigned by the investigator. Treatment determination will be made prior to study enrollment.
  Magnetic Resonance Imaging (MRI) Assessments: MRI scans will include a routine clinical MRI series.
- Stereotactic Radiation Therapy: Patients with brain metastases receiving fractionated (spread out over time) Stereotactic Radiation Therapy (FSRT). This intervention has not been assigned by the investigator. Treatment is decided prior to enrollment.
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery (SRS) | Whole Brain Radiation Therapy | Stereotactic Radiation Therapy
Started | 14 | 35 | 3
Completed | 9 | 21 | 0
Not Completed | 5 | 14 | 3
Not completed — Death | 1 | 5 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Protocol Violation | 2 | 6 | 0
Not completed — Alternate Treatment Given | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stereotactic Radiosurgery (SRS) | Whole Brain Radiation Therapy | Total
Number analyzed (Participants) | 9 | 21 | 30
Age, Continuous [Median (Full Range); unit: years] | 51 [37 to 72] | 58 [40 to 74] | 55.5 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 2 | 10 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of the Gross Tumor Volume With a BTB Opening of Ktrans > 0.005 Min-1
Description: Fifty metastatic lesions from 21 patients received WBRT and 14 lesions from 9 patients treated by SRS were analyzed. Permeability of BTB (Blood-Tumor-Barrier) was quantified by the transfer constant, Ktrans, derived from dynamic contrast enhanced (DCE)-MRI that were acquired pre, 1-2 weeks after starting, and 1-month post-radiotherapy. A percentage volume of the BM with Ktrans >0.005 min-1 (%Vall) was used to evaluate the extent of BTB opening pre-RT and subsequent changes after receiving radiotherapy. The 50 lesions, from the 21 patients treated with Whole Brain Radiation Therapy, were divided into two subgroups: low-leaky (%Vall <50%) and high-leaky, based upon pre-RT measurements. Of the 50 lesions, 7 were classified as low leaky and 43 were classified as high leaky. All 14 SRS lesions were classified as high leaky.
Time Frame: Pre-Treatment, 1-2 Weeks Post Treatment (SRS), 1 Month Post Treatment
Population: Fifty metastatic lesions from 21 patients received WBRT and 14 lesions from 9 patients treated by SRS were analyzed. All lesions were classified as high or low leaky dependent upon pre-RT permeability values.
Measure: Mean (Standard Error); unit: percentage of gross tumor volume
Units Other Than Participants: lesions
Groups:
- Stereotactic Radiosurgery (SRS): Patients with brain metastases receiving single fraction Stereotactic Radiosurgery (SRS). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed prior to SRS, at 1-2 weeks post SRS, and 1 month after SRS. The MRI scan will include a routine clinical MRI series.
  Single Fraction Stereotactic Radiosurgery (SRS): Intervention will not be assigned by the investigator. Treatment determination will be made prior to study enrollment.
  Magnetic Resonance Imaging (MRI) Assessments: MRI scans will include a routine clinical MRI series.
- Whole Brain Radiation Therapy (High Leaky Lesions): 43 Lesions from 21 Patients were highly leaky.
  Participants with brain metastases receiving fractionated (spread out over time) Whole Brain Radiation Therapy (WBRT). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed prior to RT, at 1-2 weeks post RT and 1 month after RT. The MRI scan will include a routine clinical MRI series.
  An in-house program developed to estimate vascular permeability voxel-by voxel was used to classify this WBRT group as " High Leaky" (more permeable) based upon their baseline MRI scan.
- Whole Brain Radiation Therapy (Low Leaky Lesions): 7 Lesions from 21 Patients were classified as low leaky.
  Participants with brain metastases receiving fractionated (spread out over time) Whole Brain Radiation Therapy (WBRT). This intervention is not assigned by the investigator. Treatment has been decided prior to study enrollment.
  MRI scans will be performed prior to RT, at 1-2 weeks post RT and 1 month after RT. The MRI scan will include a routine clinical MRI series.
  An in-house program developed to estimate vascular permeability voxel-by voxel was used to classify this WBRT group as " High Leaky" (more permeable) based upon their baseline MRI scan.
Arm/Group | Stereotactic Radiosurgery (SRS) | Whole Brain Radiation Therapy (High Leaky Lesions) | Whole Brain Radiation Therapy (Low Leaky Lesions)
Number analyzed (Participants) | 9 | 21 | 21
Number analyzed (lesions) | 14 | 43 | 7
percentage of gross tumor volume
  Pre-RT | 78.6 (7.4) | 85.6 (2.1) | 6.4 (3.1)
  1-2 Weeks Post RT | 74.4 (8.4) | 81.3 (2.5) | 30.2 (13.1)
  1 Month Post RT | 75.3 (5.8) | 76.7 (4.1) | 52.6 (13.5)

2. Primary Outcome: Change in Magnitude and Regional Variability of Blood Tumor Barrier (BTB)/Blood Brain Barrier (BBB) Permeability (Per Minute) in Tumor, Tumor Margin, Normal Brain and Brain Metastases
Description: An in-house program, based on a general kinetic model, along with an MRI contrast agent, Gadopentetic Acid (Gd-DTPA), will be used to estimate vascular permeability (per minute).
Time Frame: Week -2 to -1, End of Treatment (WBRT), 1-2 Weeks Post Treatment (SRS), 1 Month Post Treatment
Reporting Status: Not Posted

3. Secondary Outcome: Change in Mean K^Trans During and After Radiation Therapy
Description: Effect of radiation dose on vascular permeability (per minute) of the Blood Tumor Barrier (BTB)/Blood Brain Barrier (BBB). Permeability of BTB was quantified by Ktrans.
Time Frame: Pre-treatment and 1 Month Post Treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Only adverse events recorded in the medical chart as related to the study MRI scan or neurocognitive testing) were collected per protocol. No Non-Serious or Serious Adverse Events were reported to the study team.
Arm/Group | Stereotactic Radiosurgery (SRS) | Whole Brain Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/21
Other Adverse Events (participants affected / at risk) | 0/9 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes